CLINICAL TRIAL: NCT06477601
Title: Impact of WS-3, Menthol, and Non-menthol Cigarettes on Cigarette Smoking and Abuse Liability Among Adult Menthol Smokers: A Pilot Investigation
Brief Title: Cooling Agent Pilot Among Adult Menthol Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 160670
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Tobacco Dependence
Keywords: tobacco
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be 20 adult current menthol smokers. Participants will be randomized to continued menthol smoking (n = 4), WS-3 synthetic cooling agent cigarette smoking (n = 8), or traditional non-menthol cigarette smoking (n = 8).
Masking Description: Participants and investigators will be blind during randomization. Participants will be randomly assigned to their arm, but once assigned, participants and investigators will know which product they have been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Continued menthol smoking (Active Comparator): Current menthol smokers will be assigned to smoke study provided menthol cigarettes.
  Interventions: Other: Assigning menthol type cigarettes
- Synthetic cooling agent cigarette smoking (Experimental): Current menthol smokers will be assigned to smoke study provided synthetic cooling agent cigarettes.
  Interventions: Other: Assigning cooling agent type cigarettes
- Traditional non-menthol cigarette smoking (Experimental): Current menthol smokers will be assigned to smoke study provided traditional non-menthol cigarettes.
  Interventions: Other: Assigning traditional tobacco type cigarettes

INTERVENTIONS:
Other: Assigning cooling agent type cigarettes — This study is intended to help understand what people who smoke menthol cigarettes would do in a scenario where the Food and Drug Administration bans menthol cigarettes but allows cooling agent cigarettes.
  Arms: Synthetic cooling agent cigarette smoking
Other: Assigning traditional tobacco type cigarettes — This comparison group is intended to help understand what people who smoke menthol cigarettes would do in a scenario where the Food and Drug Administration bans menthol and cooling agent cigarettes.
  Arms: Traditional non-menthol cigarette smoking
Other: Assigning menthol type cigarettes — This comparison group is for where the Food and Drug Administration does not ban menthol cigarettes.
  Arms: Continued menthol smoking

SUMMARY:
Recent studies and market monitoring have shown that in places where menthol cigarettes are no longer available, tobacco companies have started marketing "non-menthol cooling cigarettes". Little is known about what current menthol smokers think of these non-menthol cooling cigarettes and how they compare to regular menthol cigarettes. By doing this study, the investigators hope to learn what menthol smokers think of these cigarettes and how they impact how menthol smokers smoke.

DETAILED DESCRIPTION:
The Food and Drug Administration has been considering a potential federal restriction on menthol as a characterizing flavor in combustible cigarettes, a policy that would likely significantly reduce tobacco related disparities among Black adults who smoke menthol cigarette. However, in states where this policy has been enacted and menthol cigarettes are off the market, the tobacco industry has circumvented the restriction by introducing new non-menthol cigarettes that include WS-3, a chemical that acts as a cooling agent but without use of menthol. Our team is interested in understanding the extent to which WS-3 undermines a potential future menthol ban and the impact on the reduction in cigarettes smoked, particularly among Black adults who smoke.

The overall objective of this application is to obtain effect sizes and establish feasibility for an upcoming R01 submission. Specific aims include: Aim1: Determine the change in total cigarettes per day (CPD) when using menthol cigarettes, WS-3 cigarettes, and traditional non-menthol cigarettes. The primary comparison is between WS-3 and traditional non-menthol cigarettes. Aim 2: Understand the comparative abuse liability during ad libitum use of menthol cigarettes, WS-3 synthetic cooling agent cigarettes, and traditional non-menthol cigarettes. The study intervention involves providing study participants, who are all adult current smokers with no intention to quit or alter their cigarette smoking, with either menthol cigarettes, WS-3 synthetic cooling agent cigarettes, or traditional non-menthol cigarettes. All study products are commercially available. Participants will report on their usual number of cigarettes per day and will be provided a commensurate amount of study cigarettes to allow them to make a complete switch to the study product for the duration of the 6 week research study.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smoker
* Smoke at least 5 cigarettes per day
* Smoke on at least 25 of the past 30 days
* Smoke menthol cigarettes for at least 1 year
* At least 21 years old
* Willing to try a product switch for 3 weeks and be followed for 6 weeks
* Willing to not use marijuana in place of the study product
* Willing to refrain from other tobacco product use for 3 weeks during the study
* Speak and understand English
* Willing to provide informed consent
* Own cell or landline phone
* Have reliable transportation
* Plan to remain in the Kansas City area for the full duration of the study (6 weeks)
* Bring pack of menthol cigarettes to W0 study visit

Exclusion Criteria:

* E-cigarette use on greater than 4 of the past 30 days
* Other tobacco product use on greater than 4 of the past 30 days
* Interested in quitting smoking (i.e., setting a quit date) in the next 30 day
* Current use of cessation medications
* Household member currently or previously enrolled in the study
* Currently pregnant
* Unable to provide informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-06-24 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Cigarette changes from baseline to week 3 | 3 weeks
  4.1 The primary study endpoint is changes in total cigarettes per day from baseline to week 3.

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Leavens, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Tobacco Treatment Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No